CLINICAL TRIAL: NCT02144870
Title: Randomized Control Trial on the Efficacy of Habit Reversal Treatment Programme in Children and Adolescents - a Comparison With Resource Activation Treatment
Brief Title: Efficacy of Psychotherapy Treatment of Children With Tics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Manfred Doepfner, Leading psychologist at the Department of Childhood and Adolescence Psychiatry, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: THICS-Study
Record Dates: First submitted 2014-04-14; First posted 2014-05-22 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Tic-Disorder
Keywords: Tic-Disorder, Tourette-Disorder, Habit Reversal Training, Resources activation
MeSH Terms: conditions — Tics; Tourette Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Habit Reversal Training (Active Comparator): At first patients get informed about Tics in general. Then the individual Tics are specified and the tic-reaction is looked at further. The Tic-Symptoms are observed and the premonitory urge is specified. For all individual tics a specific reversal movement is developed. Relaxation methods are introduced.
  Interventions: Behavioral: Habit Reversal Training
- Resources activation (Active Comparator): At first patients get informed about Tics in general. Through different exercises existing resources and skills are activated and strengthened. Feeling of self-esteem and self-respect are strengthened. Also the emotional awareness is strengthened. Relaxation methods are also introduced.
  Interventions: Behavioral: Resources activation

INTERVENTIONS:
Behavioral: Habit Reversal Training — awareness training, competing response training
  Arms: Habit Reversal Training
Behavioral: Resources activation
  Arms: Resources activation

SUMMARY:
The main purpose of this study is to evaluate the efficacy of a habit reversal based treatment programme compared to an alternative treatment which aims at the activation of resources in children and adolescents aged 8 to 18 years with tic disorders.

DETAILED DESCRIPTION:
The main purpose of this study is to evaluate the efficacy of a habit reversal based treatment programme (THICS, Woitecki & Döpfner, 2014) compared to an intervention aimed at the activation of resources (STARK, Perri et al., 2014) for children and adolescents with tic disorders. This habit reversal treatment programme was developed at the Department of Child and Adolescent Psychiatry and Psychotherapy at the University of Cologne and has already been evaluated in a pilot-study (Woitecki & Döpfner, 2011, 2012). The activation of resources treatment programme was also developed at this Department and is currently evaluated in different studies. Effects are expected in both interventions, but a larger effect is expected in the THICS treatment

ELIGIBILITY:
Inclusion Criteria:

* 8-18 years
* Diagnosis of chronic motor or vocal Tic (F95.1) or Tourette-Syndrome (F95.2)
* YGTSS total score F95.2>13, F95.1>9
* Tics are the main problems
* Intelligence IQ>80
* If medication, then has been stable for at least one months in medicated patients
* No change in medication treatment is planned
* Ability to participate in weekly outpatient treatment
* Acceptance of randomization

Exclusion Criteria:

Diagnosis of Autism Spectrum Disorder or Psychosis Parallel continuous psychotherapy of tics or comorbid -

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-11; Primary Completion 2017-07 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Symptom Checklist for Tic-Symptoms (FBB-TIC, parent rating) at week 8, 16 and 24 | eight weeks (T1), sixteen weeks (T2) and 24 weeks (T3)
  The FBB-TIC is used to assess Tic-Symptoms according to DSM-IV and ICD-10 rated by parents
Change in Quality of Life (Tic-HRQoL-FBB)(parent rating) | eight weeks (T1) and twenty-four weeks (T3)
  The Tic-HRQoL-FBB is used to assess impairment and quality of life through tic symptoms and other comorbid symptoms rated by parents

SECONDARY OUTCOMES:
Change in Symptom Checklist for Tic-Symptoms (FBB-/SBB-TIC), Teacher-/self-rating | eight weeks (T1), sixteen weeks (T2) and 24 weeks (T3)
  The SBB-TIC is used to assess Tic-Symptoms according to DSM-IV and ICD-10 rated by parents
Change in Symptom Checklist for Tic-Symptoms, clinical rating | eight weeks (T1), sixteen weeks (T2) and 24 weeks (T3)
  The Checklist is used to assess Tic-Symptoms according to DSM-IV and ICD-10 rated by clinicians
Change of comorbid ADHD Symptoms (FBB/SBB-ADHD), parent, teacher and self-rating | eight weeks (T1), and 24 weeks (T3)
  The Symptom Checklist for Attention Deficit/Hyperactivity Disorder (FBB-/SBB-ADHS) assess all symptom criteria according to DSM IV and ICD-10.
Change of comorbid OCD Symptoms (ZWIK-E), parent-rating | eight weeks (T1), and 24 weeks (T3)
  The ZWIK assess OCD criteria.
Change of comorbid Symptoms (CBCL/TRF/YSR), parent-/teacher-/self-rating | eight weeks (T1), and 24 weeks (T3)
  The CBCL, TRF and YSR assess a variation of different criteria.
Change in self-esteem (Harter-Scale-SBB)(self rating) | eight weeks (T1), and 24 weeks (T3)
  The Harter-Scale is used to assess self-esteem
Change in Tic-Symptoms (YGTSS-TIC), overall score | eight weeks (T1), sixteen weeks (T2) and 24 weeks (T3)
  The YGTSS is used to assess Tic-Symptoms in a semi structured interview with parents and patients
Change in Tic-Symptoms (observation) | 24 weeks (weekly assessment)
  Tic symptoms are observed through video tapes and are rated through clinicians.

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Döpfner, Prof. Dr., Study Director — Department of Childhood and Adolescent Psychiatry and Psychotherapy
Locations (1):
- University Hospital of Cologne, Department of Childhood and Adolescent Psychiatry and Psychotherapy, Cologne, Germany